CLINICAL TRIAL: NCT05611398
Title: Analysis of Lactate Monitoring Requirement in Emergent Surgical Interventions in Noncritical Traumatic Long Bone Fractures
Brief Title: Lactate Monitoring in Traumatic Long Bone Fractures Requiring Emergent Surgical Intervention
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-51
Record Dates: First submitted 2022-10-26; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Lactate Blood Increase; Trauma Blunt; Trauma, Secondary; Injury Traumatic
MeSH Terms: conditions — Hyperlactatemia; Wounds, Nonpenetrating; Compassion Fatigue; Wounds and Injuries | interventions — Orthopedic Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lactate Level Under 2 mmol/L: Patients with a lactate level below 2
  Interventions: Procedure: Orthopedic Surgery
- Lactate Level Over 2 mmol/L: Patients with a lactate level above 2
  Interventions: Procedure: Orthopedic Surgery

INTERVENTIONS:
Procedure: Orthopedic Surgery — A complete retrospective chart review was performed for all the patients' records and included all patients aged 18 years or higher who presented to Arrowhead Regional Medical Center with long bone fractures with Injury Severity Score <16 and their repair and lactate levels at the time of surgery

SUMMARY:
Serum lactate has been utilized as a standard in guiding management of orthopedic injuries. Elevated preoperative lactate has been associated with a higher likelihood of postoperative complications. However, lactate's role in guiding operative timing in non-critical long-bone fractures has not been previously explored. This study investigates lactate's role in guiding surgical timing and predicting complications secondary to delayed definitive correction in non-critical long-bone fractures with Injury Severity Score <16.

DETAILED DESCRIPTION:
Trauma is among the leading causes of death, disability, and hospitalizations each year worldwide. The majority of traumatic injuries are orthopedic in nature, making up nearly one million hospital encounters each year. According to the Center for Disease Control and Prevention, fractures are among the top 20 first-line diagnosis presenting to the emergency department. In recent years, the epidemiology of long bone fractures has been changing, with an increased incidence of fragility fractures in the elderly and high energy injuries affecting young adults. Fall-related fractures account for 61% of emergency orthopedic surgical procedures. Management of these orthopedic fractures is complex, and certain predictors such as lactate have been suggested to play a role in outcomes.

In the setting of trauma, the metabolic response of insufficient tissue perfusion is anaerobic glycolysis, with serum lactate as the final byproduct. Serum lactate serves as a circulating biomarker for organ oxygen supply and demand mismatch and is often used as a surrogate for tissue hypoxia. Normal blood lactate levels range from 0.5 to 2.2 mmol/L, with some variability in the upper limitation. Studies show early lactate clearance may be an important and independent prognostic variable in guiding management protocol for the resuscitation of trauma patients. Furthermore, several studies have presented more evidence that lactate levels can be considered a sensitive marker for patients in shock and during resuscitation with strong correlation with morbidity and mortality levels.

The goal of this study is to further investigate the role of serum lactate levels in guiding surgical timing and complications resulting from delay to the definitive surgical intervention in noncritical, traumatic patients with sustained long bone fractures.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or higher with long bone fractures with Injury Severity Score <16

Exclusion Criteria:

* Non-long bone fracture surgeries performed within the first 72 hours
* Patients who underwent external fixation prior to surgery
* Patients with inconsistent or incomplete chart data Patients with polytrauma and life-threatening injuries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was completed at the Arrowhead Regional Medical Center (ARMC) in San Bernardino County, California. The ARMC is a 456-bed acute-care teaching facility and ACS-verified level I trauma center. The ARMC emergency department (ED) is one of the busiest in the state of California with more than 100,000 visits and over 3,000 adult trauma cases annually.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Preoperative lactate levels | The estimated period of time over which preoperative lactate levels are measured occur in the initial 2 hours aft
  Preoperative lactate levels were defined as the first measured lactate level on admission of an individual who presented as a trauma patient.
Time to surgery from admission | Time to surgery from admission in the hospital is defined as the event until initial orthopedic surgery occurred after admission. The time frame of measurement was 28 days until the event occurred.
  The time that elapsed from admission to the hospital until surgery occurred
Intraoperative complications | 28 days
  Incidence of known adverse events associated with orthopedic operation
Length of total hospital stay | Length of total hospital stay from admission in the hospital is defined as the time frame between admission and discharge. The time frame of collection until the event occurred was 180 days.
  The time spent hospitalized in days.
Discharge disposition | Time frame of collection until the event occurred was 180 days.
  Once discharge was initiated did the individual get discharged home, skilled nursing facility, acute care facility.

CONTACTS AND LOCATIONS:
Overall Officials: Aldin Malkoc, MD, Study Chair — Arrowhead Regional Medical Center; Michael Neeki, DO, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarman MP, Weaver MJ, Haider AH, Salim A, Harris MB. The National Burden of Orthopedic Injury: Cross-Sectional Estimates for Trauma System Planning and Optimization. J Surg Res. 2020 May;249:197-204. doi: 10.1016/j.jss.2019.12.023. Epub 2020 Jan 25. PMID 31991329
- [Background] Frouzan A, Masoumi K, Delirroyfard A, Mazdaie B, Bagherzadegan E. Diagnostic accuracy of ultrasound in upper and lower extremity long bone fractures of emergency department trauma patients. Electron Physician. 2017 Aug 1;9(8):5092-5097. doi: 10.19082/5092. eCollection 2017 Aug. PMID 28979747
- [Background] Ekegren CL, Edwards ER, de Steiger R, Gabbe BJ. Incidence, Costs and Predictors of Non-Union, Delayed Union and Mal-Union Following Long Bone Fracture. Int J Environ Res Public Health. 2018 Dec 13;15(12):2845. doi: 10.3390/ijerph15122845. PMID 30551632
- [Background] Bakker J, Gris P, Coffernils M, Kahn RJ, Vincent JL. Serial blood lactate levels can predict the development of multiple organ failure following septic shock. Am J Surg. 1996 Feb;171(2):221-6. doi: 10.1016/S0002-9610(97)89552-9. PMID 8619454